CLINICAL TRIAL: NCT04610138
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of ZnAg Liquid Solution to Treat COVID-19 in Acutely Symptomatic Non-Hospitalized Participants
Brief Title: Study of ZnAg Liquid Solution to Treat COVID-19 Symptomatic Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clene Nanomedicine (Industry)
Collaborators: ICL Pharma (Unknown); Azidus Brazil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNMZnAg.202
Record Dates: First submitted 2020-10-28; First posted 2020-10-30 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: SARS-CoV-2; COVID; COVID-19; Corona Virus
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:2 to receive ZnAg (low dose): ZnAg (high dose) placebo in a double-blind fashion in addition to standard supportive care. Within the active treatment arm, participants will be randomized to receive either low or high dose ZnAg.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, investigators, and coordinators will be blinded to the investigational product. The study data will remain blinded until database lock and authorization of data release according to standard operating procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active treatment with 60 ml low-dose ZnAg (Experimental): (Zn 6 ug/ml and Ag 10 ug/ml; equivalent to 0.6 mg Ag, 0.36 mg Zn), po q12 hours
  Interventions: Drug: CNM-ZnAg
- Active treatment with 60 ml high-dose ZnAg (Experimental): (Zn 12 ug/ml and Ag 20 ug/ml; equivalent to 1.2 mg Ag, 0.72 mg Zn), po q12 hours;
  Interventions: Drug: CNM-ZnAg
- 60 ml matching placebo (Placebo Comparator): 60 ml matching placebo, po q12 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNM-ZnAg — ZnAg liquid solution
  Arms: Active treatment with 60 ml high-dose ZnAg; Active treatment with 60 ml low-dose ZnAg
Drug: Placebo — Water
  Arms: 60 ml matching placebo

SUMMARY:
This is a multi-site, randomized, double-blind, placebo-controlled study assessing the efficacy and safety of ZnAg liquid solution in symptomatic participants with acute COVID-19 that are not hospitalized at the time of enrollment.

DETAILED DESCRIPTION:
This is a multi-site, randomized, double-blind, placebo-controlled study assessing the efficacy and safety of ZnAg liquid solution in symptomatic participants with acute COVID-19 (PCR documented SARS-CoV-2 infection) that are not hospitalized at the time of enrollment (e.g., present to an emergency room without being admitted to the hospital or diagnosed in an outpatient clinic setting).

Participants must have presented with two or more symptoms of acute COVID-19 (within 96 hours prior to the Baseline visit) self-reported as moderate or severe at the Baseline visit, including fever, myalgia, fatigue, chest tightness, chills, cough, diarrhea, gastrointestinal distress, headache, sore throat, congestion or runny nose, ageusia, anosmia, nausea, tingling or numbness in the extremities, or shortness of breath. SARS-CoV-2 infection must be confirmed by polymerase chain reaction (PCR) testing within 96 hours prior to the Baseline visit.

Participants who meet all inclusion criteria and none of the exclusion criteria and who formally consent to participate will be randomized 1:1:2 to receive ZnAg (low dose) : ZnAg (high dose) placebo in a double-blind fashion in addition to standard supportive care. Within the active treatment arm, participants will be randomized to receive either low or high dose ZnAg.

* Active treatment with 60 ml low-dose ZnAg (Zn 6 ug/ml and Ag 10 ug/ml; equivalent to 0.6 mg Ag, 0.36 mg Zn), po q12 hours or;
* Active treatment with 60 ml high-dose ZnAg (Zn 12 ug/ml and Ag 20 ug/ml; equivalent to 1.2 mg Ag, 0.72 mg Zn), po q12 hours;
* 60 ml matching placebo, po q12 hours

Participants who become clinically unstable during the course of the study (e.g., requiring high-flow supplemental oxygen or mechanical ventilatory support) per the judgement of the site investigator will be admitted to a hospital and their clinical status (e.g., vital status, hospitalization status, respiratory status, COVID-19 ordinal scale) will continue to be tracked per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 40 - 90 years (inclusive)
2. Acute onset (within 96 hours of the Baseline visit) of two or more COVID-19 symptoms self-rated as moderate-to-severe, including fever, myalgia, fatigue, chest tightness, chills, cough, diarrhea, gastrointestinal distress, headache, sore throat, congestion, or runny nose, ageusia, anosmia, nausea, tingling or numbness in the extremities, or shortness of breath.
3. Laboratory-confirmed SARS-CoV-2 infection as determined by positive PCR in a sample collected ≤ 96 hours prior to the Baseline visit.
4. PGI-Severity and CGI-Severity assessments of 'Mild', 'Moderate, or 'Severe' at the Screening visit (e.g., cannot be 'Normal').
5. Participant (or legally authorized representatives) provides informed consent prior to the initiation of any study procedures.
6. Participant is willing and able to follow all study procedures and assessments according to the study protocol.
7. Participant is able to consume 60 ml of fluid orally twice daily.
8. Women of childbearing potential must agree to either abstinence or use at least one primary form of contraception, not including hormonal contraception from the time of screening through the end of study.

Exclusion Criteria:

1. Unable or unwilling to take ZnAg liquid solution or matching placebo as directed.
2. Hospitalized prior to Baseline for COVID-19 management.
3. Need for hospitalization and/or ventilatory support at Baseline.
4. The emergence of any disease during study, other than COVID-19 that could better explain the participants' signs and symptoms.
5. Severe disease: respiratory distress, or requiring supplemental oxygen, or SpO2 ≤ 93% on room air, or tachypnea (respiratory rate ≥ 30 breaths/min) at Baseline.
6. History or presence of serious or acute heart disease such as uncontrolled cardiac dysrhythmia or arrhythmia, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure (NYHA class 3 or 4).
7. Legal incapacity or limited legal capacity.
8. Women of childbearing potential who do not agree to use either abstinence or at least one primary form of contraception, not including hormonal contraception from the time of screening through the end of the study.
9. Pregnant or breastfeeding.
10. Participation in another clinical study with an investigational product within the prior 12 months (per Resolution 251/1997).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Time to substantial alleviation of COVID-19 symptoms. | Up to 28 days.
  Time to substantial alleviation of COVID-19 symptoms up to 28-days, over a continuous period ≥ 48 hours (confirmed symptom resolution), defined as PGI-Severity of 'Normal' in Participants whose Baseline PGI-Severity value was 'Mild'; or, a PGI-Severity of 'Normal' or 'Mild' in participants whose Baseline PGI-Severity value was 'Moderate' or 'Severe'.

SECONDARY OUTCOMES:
Time to complete alleviation of COVID-19 symptoms. | Up to 28 days.
  Time to complete alleviation of COVID-19 symptoms up to 28- days, over a continuous period ≥ 48 hours (confirmed symptom resolution).
Proportion of participants who are hospitalized, requires hospitalization or are deceased. | Up to 28 days
  Proportion of participants who are hospitalized, require hospitalization, or are deceased from Baseline to Day 28. Hospitalization will be determined by Investigator's clinical judgement. Where applicable, Investigators should follow local recommendations for hospitalization of patients with COVID-19 within their institution.

OTHER OUTCOMES:
Number of alive hospital free days at Day 28. | 28 days
  Days from baseline participant remains alive.
Mean change from Baseline to Day 8, Day 14, Day 21, and Day 28 in SARS-CoV-2 viral load. | Up to 28 days
  Mean change from Baseline to Day 8, Day 14, Day 21, and Day 28 in SARS-CoV-2 viral load (Cycle Thresholds, Ct) , and time to non-detectable virus levels assessed by RT-qPCR.
Change from Baseline to Day 8, Day 14, Day 21, and 28 in the slope of oxygen saturation levels (SpO2) assessed per protocol. | up to 28 days
  Oxygen saturation will be obtained after the participant has been resting for 5 minutes.
Clinical Global Impression (CGI) Severity and Change measures from Baseline to Day 8, Day 14, Day 21, and 28. | Up to 28 days
  Measured by changes in participant rated Clinical Global Impression.
Patient Global Impression (PGI) Severity and Change measures from Baseline to Day 8, Day 14, Day 21, and 28. | Up to 28 days
  Measured by changes in participant rated Patient Global Impression.
Change in the area under the curve for Net Symptom Burden from Baseline to Day 8, Day 14, Day 21, and 28. | Up to 28 days
  Summary measure integrating semi-daily serial assessments of a subject's symptom count and severity over the duration of the study.
Change in clinical status from Baseline to Day 8, Day 14, Day 21, and Day 28. | Up to 28 days
  Assessed by the Clinical Status Ordinal Scale established in the remdesivir ACTT study. Scale is 1-8, with 1 being the least severe and 8 being the most severe (death).
All-cause mortality rate at Day 28. | 28 days
  Rate of deceased participants at day 28.
Proportion of subjects who have not returned to "normal" at the day 21 and day 28 visits. | 28 days
  Proportion of subjects who do not have a PGI-Severity or CGI-Severity assessment of "normal" at the day 21 and day 28 visits.

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - PROCAPE, Santo Amaro, Recife
  - Projeto Praca Onze, Centro, Rio de Janeiro
  - IBPClin, Glória, Rio de Janeiro
  - Casa de Saúde, Campinas, Sau Paulo
  - IPECC, São Paulo, State of Sau Paulo

IPD SHARING:
Plan to Share IPD: No